CLINICAL TRIAL: NCT00607334
Title: Experimental Word Learning in Children With Normal Development and Children With Language Impairment
Brief Title: Experimental Word Learning in Children With and Without Language Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Debora Maria Befi-Lopes, University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24061316
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2007-10

CONDITIONS: Developmental Language Disorders
Keywords: Child Language; Language Therapy; Vocabulary
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GP (Experimental): Children with Developmental Language Impairments were enrolled in this group.
  Interventions: Behavioral: Word-learning
- GC (Experimental): Children with normal language development were enrolled in this group.
  Interventions: Behavioral: Word-learning

INTERVENTIONS:
Behavioral: Word-learning — Exposure to five nonwords for three sessions of controlled interaction with the experimenter
  Arms: GP
Behavioral: Word-learning — Exposure to five nonwords for three sessions of controlled interaction with the experimenter
  Arms: GC

SUMMARY:
The purpose of this study is to compare the performances of normally developing children and children with Language Impairment (LI) in three different experimental settings designed to promote vocabulary acquisition. This comparison will also provide evidence to support different intervention approaches designed to increase vocabulary abilities, which has been proved to be one of the major deficits of young children with LI.

ELIGIBILITY:
Inclusion Criteria:

* For GP subjects: - diagnosis of Language Impairment
* enrolled in language therapy
* age between 3:0 (years:months) and 3:11
* For GC subjects: - normal performance in a language screening procedure
* normal performance in an expressive vocabulary test

Exclusion Criteria:

* For GP subjects: - hearing impairments
* diagnosed neurological or behavioral conditions
* major cognitive impairment
* For GC subjects: - communication complaints from caregivers
* history of previous enrollment in language therapy

Ages: 36 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2003-07; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Performance on a post-test administered after every word-learning session. | Three weeks

SECONDARY OUTCOMES:
Occurence of correct spontaneous productions of the taught words during the experimental procedure | Three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debora M. Befi-Lopes, PhD, Study Chair — University of Sao Paulo; Juliana P. Gândara, PhD student, Principal Investigator — University of Sao Paulo
Locations (1):
- USP - Faculty of Medicine - Department of Physiotherapy, Communication Sciences and Disorders, Occupational Therapy, São Paulo, São Paulo, Brazil